CLINICAL TRIAL: NCT00441597
Title: Does Atorvastatin Reduce Ischemia-Reperfusion Injury in Humans in-Vivo?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: G Rongen, dept Pharmacology Toxicology UMCN
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: atorv01
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Ischemia Reperfusion Injury; Cardiovascular Disease
Keywords: ischemia reperfusion injury; atorvastatine; preconditioning; cardiovascular disease
MeSH Terms: conditions — Reperfusion Injury; Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): first 3 day treatment placebo and 4 weeks later three day treatment with atorvastatin 80 mg
  Interventions: Drug: atorvastatin
- 2 (Active Comparator): first 3 day treatment atorvastatin 80 mg and 4 weeks later three day treatment with placebo
  Interventions: Drug: atorvastatin
- 3 (No Intervention): 3 days treatment with placebo twice

INTERVENTIONS:
Drug: atorvastatin — atorvastatine 80mg, during 3 days
  Other Names: lipitor
  Arms: 1; 2

SUMMARY:
To study the impact of 3 day exposure to atorvastatin 80mg on Annexin A5 targeting after ischemic exercise in the non-dominant forearm.

DETAILED DESCRIPTION:
3-Hydroxy-3-methylglutaryl coenzyme A reductase inhibitors (also known as statins) have been found to reduce cardiovascular events. This protective effect has been traditionally explained by lowering plasma cholesterol and subsequent reduced progression of atherosclerosis. However in animal experiments statins have also shown the ability to induce pharmacologic preconditioning and thereby reduce infarct size. This effect contributes to the beneficial effect of statins on reducing of cardiovascular events. In order to differentiate between these two mechanisms of protection we will study the effect of atorvastatin on ischemia reperfusion damage after a short exposure to atorvastatin, before the lipid lowering effect of atorvastatin becomes apparent.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-50 years
* Informed consent
* Physical able to perform ischemic exercise

Exclusion Criteria:

* History of any cardiovascular disease
* Hypertension (in supine position: systole > 140 mmHg, diastole > 90 mmHg)
* Diabetes mellitus (fasting glucose > 7.0 mmol/L or random glucose > 11.0 mmol/L)
* Hyperlipidaemia (fasting total cholesterol > 5.5 mmol/l)
* Alanine-Amino-Transferase (ALAT) >90 U/L
* Creatinine Kinase (CK) >440 U/L
* Drug or alcohol abuse
* Concommitant chronic use of medication
* Administration of radioactivity in research setting during the last 5 years
* Participation to any drug-investigation during the previous 60 days as checked with VIP check according to CRCN standard procedures

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Annexin A 5 targeting in the non dominant thenar muscle after ischemic exercise, as a indicator for ischemia reperfusion injury. | 60 and 240 minutes after ischemic exercise

SECONDARY OUTCOMES:
workload during ischemic exercise | workload during 10minutes of ischemic exercise
effect of 3-day treatment with atorvastatin 80mg daily on serum lipid levels | fasting lipid levels before and at first day after 3 day treatment with atorvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD PhD, Principal Investigator — RUMCN
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546
- [Background] Riksen NP, Smits P, Rongen GA. Ischaemic preconditioning: from molecular characterisation to clinical application--part II. Neth J Med. 2004 Dec;62(11):409-23. PMID 15685892